CLINICAL TRIAL: NCT04294407
Title: Assessment of Upper Extremity Muscle Spasticity and Impedance Using the Movement and Electromyographical Analyses
Brief Title: Using the Movement and Electromyographical Analyses to Assess the Muscle Spasticity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-107-317
Record Dates: First submitted 2020-01-07; First posted 2020-03-04 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: spasticity; Modified Ashworth Scale (MAS); electromyography; kinetics; impedance
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke group: 20 to 65 years old patients, with the clinical diagnosis of stroke (Mini-mental state examination (MMSE) score of ≥25)
  Interventions: Other: No intervention
- Healthy group: 20 to 65 years old healthy subjects, without the clinical diagnosis of stroke
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention in this study

SUMMARY:
This study intends to use an dynamometer and surface electromyography to objectively and quantitatively measure the corresponding force and electromyography signal generated when the hand joint receives stretching by doing circular motion, and further explore the differences and relationships of existing muscle spasm classification, kinetic and kinematic data, upper extremity performance, activity of daily life. In addition, to investigate the differences of kinetic and kinematic data between stroke patient and healthy participants during doing hand circular motion activity.

DETAILED DESCRIPTION:
Purpose 1 : To collect upper limb muscle activity parameters of healthy adults and stroke patients to establish a database of doing hand circular motion activity.

Purpose 2 : To test the reliability of this refined muscle testing by collecting the muscle activity during hand circular motion activity.

Purpose 3 : To compare the results of the EMG signal strength with other evaluation methods such as the modified Ashworth scale and dynamometer to understand the relationship between the EMG signal and each evaluation results.

Purpose 4 : To compare the differences in electromyographic signals, muscle strength, and joint angle between healthy adults and stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 65 years old
* with the clinical diagnosis of stroke
* Mini-mental state examination (MMSE) score ≥ 25 points

Exclusion Criteria:

* pain, subluxation or related medical history of shoulder, elbow, and wrist joints within six months
* surgery on shoulder, elbow or wrist
* with muscle or nerve disorders or diseases that significantly affect the performance of the upper extremities

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with stroke will be recruited from the Department of Rehabilitation in National Cheng Kung University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Surface electromyography device--Baseline | Baseline
  The wireless EMG system will be used to record muscle activity of biceps brachii, triceps brachii, anterior deltoid, and brachioradialis during the hand circular motion activity. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Surface electromyography device--3 days after baseline | 3 days after baseline
  The wireless EMG system will be used to record muscle activity of biceps brachii, triceps brachii, anterior deltoid, and brachioradialis during the hand circular motion activity. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Surface electromyography device--6 days after baseline | 6 days after baseline
  The wireless EMG system will be used to record muscle activity of biceps brachii, triceps brachii, anterior deltoid, and brachioradialis during the hand circular motion activity. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Dynamometer device- muscle strength--Baseline | Baseline
  A digital dynamometer will be used to measure the maximum elbow flexion/extension force as muscle strength. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Dynamometer device- range of motion--Baseline | Baseline
  A digital dynamometer will be used to measure the range of motion of elbow flexion/extension. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Dynamometer device- muscle strength--3 days after baseline | 3 days after baseline
  A digital dynamometer will be used to measure the maximum elbow flexion/extension force as muscle strength. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Dynamometer device- range of motion--3 days after baseline | 3 days after baseline
  A digital dynamometer will be used to measure the range of motion of elbow flexion/extension. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Dynamometer device- muscle strength--6 days after baseline | 6 days after baseline
  A digital dynamometer will be used to measure the maximum elbow flexion/extension force as muscle strength. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Dynamometer device- range of motion--6 days after baseline | 6 days after baseline
  A digital dynamometer will be used to measure the range of motion of elbow flexion/extension. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Modified Ashworth Scale--Baseline | Baseline
  Modified Ashworth Scale (MAS) is a useful assessment tool to classify spasticity.The testing procedure of the MAS is to passively move the joint by the examiner and to feel the resistance during the movements. The scoring of the MAS included 6 level (0, 1, 1+, 2, 3, 4), where no increase muscle tone was score as 0 and rigid joint was score as 4. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Modified Ashworth Scale--3 days after baseline | 3 days after baseline
  Modified Ashworth Scale (MAS) is a useful assessment tool to classify spasticity.The testing procedure of the MAS is to passively move the joint by the examiner and to feel the resistance during the movements. The scoring of the MAS included 6 level (0, 1, 1+, 2, 3, 4), where no increase muscle tone was score as 0 and rigid joint was score as 4. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)
Modified Ashworth Scale--6 days after baseline | 6 days after baseline
  Modified Ashworth Scale (MAS) is a useful assessment tool to classify spasticity.The testing procedure of the MAS is to passively move the joint by the examiner and to feel the resistance during the movements. The scoring of the MAS included 6 level (0, 1, 1+, 2, 3, 4), where no increase muscle tone was score as 0 and rigid joint was score as 4. These data would be collected three times. (Baseline, 3 days after baseline, 6 days after baseline)

SECONDARY OUTCOMES:
The Fugl-Meyer Upper Extremity Scale | Baseline
  The Fugl-Meyer Upper Extremity Scale is an assessment scale for upper limb function of stroke patients. The scale has 33 movements, which can be rated as 0 to 2 points, of which 0 is impossible and 1 is achievable. 2 points can be completely achieved. FMUE scale has good reliability and validity.
Box and Block Test | Baseline
  The main purpose of the BBT test is to measure the function of the hand. The test method is to calculate the number of blocks that can be moved from one side of the box across the partition to the other side with one hand in one minute.
Action Research Arm Test | Baseline
  ARAT is a tool used to evaluate the function of upper limbs of stroke patients. The main test content is to reach out and grasp different objects in a standardized environment, and score the action based on the time to complete the action. There are 19 test items, each of which is scored 4 levels (0 ~ 3). The higher the score, the better the movement performance.
Motor Activity Log | Baseline
  It is mainly used to evaluate daily life functions, including the frequency of use of motion and the evaluation of motion quality. It is a five-point questionnaire with a total of about 30 questions. The average score of the two items of frequency of use and motion quality will be calculated separately.
EQ-5D | Baseline
  It is mainly used to assess the quality of life. It is a questionnaire-type scale with a total of six questions. Check the descriptions that match your condition (for example, I cannot perform my daily activities) and score my health status today. 0 to 100 points (100 points: best state; 0 points: worst state of health)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan